CLINICAL TRIAL: NCT01970358
Title: A Phase I Study With a Personalized NeoAntigen Cancer Vaccine in Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Ott, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Patrick Ott, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-240
Record Dates: First submitted 2013-10-09; First posted 2013-10-28 (Estimated); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Melanoma; Melanoma vaccine; Adjuvant therapy
MeSH Terms: conditions — Melanoma | interventions — poly ICLC; Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Personalized NeoAntigen Cancer Vaccine (Experimental): - NeoVax (peptides + poly-ICLC)
  Poly-ICLC: 4 x 0.5 mg (total dose 2 mg) given on days Days 1, 4, 8, 15, 22, 78, and 134
  Peptides: 4 x 300 mcg per peptide given on days Days 1, 4, 8, 15, 22, 78, and 134
  Interventions: Biological: Poly-ICLC; Biological: Peptides

INTERVENTIONS:
Biological: Poly-ICLC
  Other Names: Hiltonol
Biological: Peptides
  Other Names: NeoAntigen peptides

SUMMARY:
This research study is evaluating a new type of melanoma vaccine called "Personalized NeoAntigen Cancer Vaccine". The purpose of this study is to determine if it is possible to make and administer safely a vaccine against melanoma by using information gained from specific characteristics of the participant's own melanoma. It is known that melanomas have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the melanoma to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

DETAILED DESCRIPTION:
The study is an open label, phase I trial in which patients with high-risk melanoma are immunized with up to 20 peptides that are both specific to the patient's tumor cells (i.e., not found in their normal cells) and unique to the patient (i.e., "personal"). These peptides are encoded by missense mutations, in-frame gene fusions and novel open reading frame mutations (collectively known as "neoantigens") that have occurred within that patient's tumor cells and are identified through DNA and RNA sequencing. Up to 20 peptides about 20-30 amino acids in length will be prepared for each patient and will be administered together with the immune adjuvant poly-ICLC. The personalized NeoAntigen Cancer Vaccine consists of peptides + poly-ICLC and is called "NeoVax." This phase 1 study is designed to demonstrate that the combination of personalized neoantigen peptides and poly-ICLC is safe, feasible, and induces strong tumor-specific T cell immunity.

The trial has a two-stage enrollment process. Eligible patients will be initially entered into the trial to undergo surgery with the intent to resect all melanoma detectable clinically and on radiographic scans. Patients will be reassessed for eligibility prior to the first vaccination and will continue onto the treatment phase of the trial if secondary eligibility criteria are met. Patients with tumors that are not completely resected and/or that provide inadequate DNA and/or RNA for sequencing will be removed from the trial and replaced. After NeoVax has been prepared, the vaccine will be administered on days 1, 4, 8, 15, and 22 (priming phase), and on days 78 and 134 (booster phase).

Five patients will be entered for the initial safety evaluation (Cohort 1). If none or only 1 patient experiences a DLT on Cohort 1, an additional 10 patients will be treated at this dose to increase the likelihood of detecting serious toxicities, to complete biologic correlative endpoints, and to gain preliminary experience with clinical tumor activity. If two or more patients in Cohort 1 experience dose limiting toxicity (DLT) during the first 7 weeks of treatment, then the dose of poly-ICLC will be reduced by 50% and 5 patients will be enrolled into Cohort -1. If none or only 1 patient experiences a DLT on Cohort -1, then an additional 10 patients will be enrolled as described above. If two or more patients in Cohort -1 experience a DLT, then the study will be stopped. If four or more patients in the expansion cohort experience dose limiting toxicity (DLT) during the first 7 weeks of treatment, then the dose expansion cohort will be determined to have unacceptable toxicity and the study will be stopped prior to completion of enrollment of the expansion cohort.

ELIGIBILITY:
Inclusion Criteria (all must be met):

* Patient is willing and able to give written informed consent.
* Patient is agreeable to allow tumor and normal tissue samples to be submitted for complete exome and transcriptome sequencing.
* Pathologically confirmed, clinically evident (by physical examination or radiographic imaging) stage IIIB, IIIC, IVM1a, or IVM1b cutaneous melanoma (anatomic stages T1-4b N1a and T1-4b N2a not included). The current diagnosis may be the patient's first diagnosis of melanoma or recurrent melanoma after previous diagnosis of an earlier stage melanoma.
* Patients will undergo complete resection of their primary melanoma (if not already removed) and all regional metastatic disease with the intent of rendering them free of melanoma.
* The patient must be free of unresectable metastatic disease within 4 weeks prior to the surgery being performed with the intention to remove all melanoma.
* This pre-surgery baseline assessment must be documented by complete physical examination and imaging studies. Imaging studies must include a total body PET-CT in conjunction with a brain MRI (or head CT if brain MRI is contraindicated). If a PET/CT scan cannot be done, a CT of the neck, chest, abdomen, and pelvis should be performed.
* Patients may have received prior interferon alpha (IFN-α), but must have discontinued IFN-α therapy within 4 weeks prior to enrollment on the trial. Patients who have not received prior adjuvant therapy should be informed of the potential therapeutic benefit of IFN-α.
* Previous radiation therapy, including after the surgical resection, is allowed as long as 14 days have elapsed between the radiation and initiation of first vaccination with NeoVax.
* Age ≥ 18 years.
* ECOG performance status of 0 or 1
* Normal organ and bone marrow function as defined below:
* Leukocytes ≥ 3,500/mcL
* Absolute lymphocyte count > 800/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Hemoglobin > 10.0 g/dL
* Total serum bilirubin < 1.0 x institutional upper limit of normal
* AST (SGOT)/ALT (SGPT) < 2.0 x institutional upper limit of normal
* Serum creatinine< 1.5 x institutional upper limit of normal
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) before entry onto the trial and within 7 days prior to start of study medication because the effects NeoVax on the developing human fetus are unknown. It is the investigator's responsibility to repeat the pregnancy test should start of treatment be delayed.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from sexual activity throughout the study, starting with visit 1 through 4 weeks after the last dose of study therapy. Approved contraceptive methods include, for example: intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
* Male patients must agree to use an adequate method of contraception starting with the first dose of NeoVax through 4 weeks after the last dose of study therapy.

Exclusion Criteria (one or more will exclude from participation):

* Prior treatment with immune-modulatory agents including, but not limited to: IL-2, CTLA-4 blockade, PD-1/PD-L1 blockade, CD40 stimulation, CD137 stimulation with the exception of INF-α given as adjuvant treatment for high-risk, surgically resected melanoma
* Prior investigational, melanoma-directed, cancer vaccine therapy
* Prior chemotherapy, including targeted therapy such as BRAF or MEK inhibition
* Treatment with other investigational products within the last 2 months prior to entry into this study
* Previous bone marrow or stem cell transplant
* Concomitant therapy with any anti-cancer agents, other investigational anti-cancer therapies, or immunosuppressive agents; chronic use of systemic corticosteroids
* Use of a non-oncology vaccine therapy for prevention of infectious diseases (up-to) 4 weeks prior to enrollment to the study. Patients may not receive any non-oncology vaccine therapy during the period of NeoVax administration and until at least 8 weeks after the last dose of study therapy
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases
* Mucosal melanoma or uveal melanoma are not allowed
* Active, known, or suspected autoimmune disease or immunosuppressive conditions with the exception of vitiligo, type 1 diabetes, residual autoimmune-related hypothyroidism requiring hormone replacement, or psoriasis not requiring systemic treatment.
* Concomitant treatment with corticosteroids greater than physiologic doses (used in the management of cancer or non-cancer-related illnesses). Topical (if not including the proposed vaccination sites) or inhalational steroids are allowed.
* Known chronic infections with HIV, hepatitis B or C
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs.
* Pregnant women are excluded from this study because personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ott, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Srikrishna D, Sachsenmeier K. We need to bring R0 < 1 to treat cancer too. Genome Med. 2021 Jul 26;13(1):120. doi: 10.1186/s13073-021-00940-9. PMID 34311780
- [Derived] Hu Z, Leet DE, Allesoe RL, Oliveira G, Li S, Luoma AM, Liu J, Forman J, Huang T, Iorgulescu JB, Holden R, Sarkizova S, Gohil SH, Redd RA, Sun J, Elagina L, Giobbie-Hurder A, Zhang W, Peter L, Ciantra Z, Rodig S, Olive O, Shetty K, Pyrdol J, Uduman M, Lee PC, Bachireddy P, Buchbinder EI, Yoon CH, Neuberg D, Pentelute BL, Hacohen N, Livak KJ, Shukla SA, Olsen LR, Barouch DH, Wucherpfennig KW, Fritsch EF, Keskin DB, Wu CJ, Ott PA. Personal neoantigen vaccines induce persistent memory T cell responses and epitope spreading in patients with melanoma. Nat Med. 2021 Mar;27(3):515-525. doi: 10.1038/s41591-020-01206-4. Epub 2021 Jan 21. PMID 33479501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: April 2014 through July 2016.
Pre-assignment Details: Participant consent/screening was conducted in two stages. Participants first had surgery with the intention to remove all melanoma. After confirmation of complete tumor resection by pathologic review and determination of adequacy of DNA and RNA from tumor tissue for sequencing, participants were reconsented for generation of the vaccine. Participants with tumors that were not completely resected and/or that provided inadequate DNA and/or RNA for sequencing were removed from the trial.
Period: Overall Study
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Started | 15
Completed | 8 (Completed all doses of NeoVax.)
Not Completed | 7
Not completed — Unable to make NeoVax or NeoVax not viable | 3
Not completed — Ineligible at time of second consent | 4

BASELINE CHARACTERISTICS:
Groups:
- Personalized NeoAntigen Cancer Vaccine: - NeoVax (peptides + poly-ICLC)
  Poly-ICLC: 4 x 0.5 mg (total dose 2 mg) given on days Days 1, 4, 8, 15, 22, 78, and 134
  Peptides: 4 x 300 mcg per peptide given on days Days 1, 4, 8, 15, 22, 78, and 134
  Poly-ICLC
  Peptides
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] — Age in years at enrollment.
  years | 61 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Melanoma AJCC Stage [Count of Participants; unit: Participants] — IIIB: Tumor with 1 positive lymph node (micrometastasis) or in-transit/satellite/microsatellite metastases without nodal involvement.
  IIIC: Tumor with multiple or macroscopic lymph node metastases, or in-transit/satellite/microsatellite metastases with regional lymph node involvement.
  IV M1a: Distant metastases to skin, subcutaneous tissue, or distant lymph nodes only.
  IV M1b: Distant metastases to the lung (may include M1a sites but no other visceral metastases).
  Lower stages (IIIB/IIIC) indicate better clinical outcomes, whereas higher stages (IV) indicate worse clinical outcomes.
  Participants
    IIIB | 3
    IIIC | 7
    IV M1a | 3
    IV M1b | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical and/or Laboratory Dose-limiting Toxicities
Description: Number of participants experiencing any of the following:
  * Grade-3 or -4 toxicity that is definitely, probably, or possibly related to the administration of vaccine
  * Grade-3 or -4 abnormal laboratory value that is definitely, probably, or possibly related to the administration of vaccine if it persists for more than 7 days, requires hospitalization, or medical intervention
  * Any grade-3 or grade- 4 toxicity that is considered, in the opinion of the investigator, to be dose-limiting
  * Any death related to study treatment A minimum of 3 vaccinations and absence of DLTs are required for a patient to complete the 7-week DLT observation period successfully.
Time Frame: 7 weeks from first study drug administration
Population: Number of participants receiving NeoVax.
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Proportion of Participants for Whom Sequencing and Analysis Leads to Identification of at Least 10 Actionable Peptides to Initiate Vaccine Production
Description: The proportion of participants for whom sequencing and analysis leads to identification of at least 10 actionable peptides to initiate vaccine production. The primary assessment of feasibility will be based on on all participants enrolled with a confirmation of completely resected tumor and with adequate DNA and RNA for sequencing. NeoVax would be feasible if no more than 50% of participants have fewer than 10 actionable peptides or have NeoVax available more than 12 weeks after confirmation of complete resection. If 4 or fewer of the first 15 participants have insufficient vaccine or first dose delays of more than 12 weeks, then the upper bound of the one-sided 90% exact confidence interval will be less than 50% and we will consider the process feasible. If 5 or more of the first 15 patients have insufficient or delayed vaccine, we will consider the vaccine not feasible. The planned vaccination regimen will be administered even if the feasibility endpoints are not met.
Time Frame: 12 weeks
Population: Number of participants with complete resection and adequate DNA/RNA for sequencing.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Number analyzed (Participants) | 11
Proportion of participants | 0.73 [0.44 to 0.92]

3. Secondary Outcome: Proportion of Participants With Specific Cellular Immune Responses Following Administration of NeoVax
Description: The induction of IFN-γ T-cell response will be based on ELISPOT assessments taken prior to vaccine administration and at week 16. The proportion of participants who achieve more than 55 SFU/10**6 PBMC or 3 times their baseline level will be presented with a 90% exact binomial confidence interval. Based on a cohort of size 15, the confidence interval will be no wider than 0.46.
Time Frame: 16 weeks
Population: Participants receiving NeoVax.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Number analyzed (Participants) | 8
Proportion of participants | 1.00 [0.69 to 1.00]

4. Secondary Outcome: Proportion of Participants Alive Without Progression at Two Years After Surgery Following Administration of NeoVax
Description: The proportion of participants alive, without disease progression at two years after resection estimated using the method of Kaplan-Meier. The endpoint is calculated as the time between pathological confirmation of complete resection and the first of disease recurrence or death. The follow-up of participants disease-free at the time of study reporting is censored at the time of the last study visit. Participants disease-free at the time of their last assessment and who have either been lost to follow-up or withdrawn consent will have their follow-up censored at the time of the last study assessment.
Time Frame: 2 Years
Population: Participants who received NeoVax.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Personalized NeoAntigen Cancer Vaccine
Number analyzed (Participants) | 8
proportion of participants | 0.75 [0.40 to 0.91]

ADVERSE EVENTS:
Time Frame: Total of 2 years after treatment initiation.
Description: Adverse events assessments every 3 months at re-staging follow-up visits (+/- 1 week) to continue until initiation of a new therapy for recurrent disease, withdrawal of consent, or death, whichever occurs first. All participants who receive one or more doses of NeoVax are included in the safety analysis.
Arm/Group | Personalized NeoAntigen Cancer Vaccine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized NeoAntigen Cancer Vaccine (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 4 (10)
Injection site reaction (General disorders) | 8 (18)
Pain (General disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Wart-Like Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT01970358/Prot_SAP_000.pdf